CLINICAL TRIAL: NCT01428622
Title: Single Dose Comparison of 3 Doses of Olodaterol in Double Fixed Dose Combination With BI54903 vs. 3 Doses of Olodaterol Mono in Free Combination
Brief Title: Olodaterol Bridging Study in Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1249.7; 2011-000935-98 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-08-25; First posted 2011-09-05 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — olodaterol

ARMS (7):
- Placebo + BI 54903 (Placebo Comparator): patient to receive 2 puffs of respimat "A" and 2 puffs of respimat "B"
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol low dose + BI54903 (Experimental): patient to receive 2 puffs of respimat "A" and 2 puffs of respimat "B"
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol medium dose + BI54903 (Active Comparator): patient to receive 2 puffs of each device
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol high dose + BI54903 (Experimental): patient to receive 2 puffs of each device
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol l dose + BI54903 (Experimental): patient to receive 2 puffs of each device
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol m dose + BI54903 (Experimental): patient to receive 2 puffs of each device
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903
- Olodaterol h dose + BI54903 (Experimental): patient to receive 2 puffs of each device
  Interventions: Device: Respimat; Drug: Olodaterol; Drug: Olodaterol & BI54903; Drug: BI54903

INTERVENTIONS:
Device: Respimat — aqueous and ethanolic solution
  Arms: Placebo + BI 54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol low dose + BI54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol medium dose + BI54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol high dose + BI54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol l dose + BI54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol m dose + BI54903
Device: Respimat — aqueous and ethanolic solution
  Arms: Olodaterol h dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Placebo + BI 54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol low dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol medium dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol high dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol l dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol m dose + BI54903
Drug: Olodaterol — aqueous solution
  Arms: Olodaterol h dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Placebo + BI 54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol low dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol medium dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol high dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol l dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol m dose + BI54903
Drug: Olodaterol & BI54903 — ethanolic solution
  Arms: Olodaterol h dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Placebo + BI 54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol low dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol medium dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol high dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol l dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol m dose + BI54903
Drug: BI54903 — ethanolic solution
  Arms: Olodaterol h dose + BI54903

SUMMARY:
The aim of the study is to establish the olodaterol dose in the ethanolic fixed dose combination (FDC) with BI 54903 which is equivalent in bronchodilator effect and systemic exposure to the 5 µg olodaterol reference dose in the aqueous inhalation solution (AIS).

ELIGIBILITY:
Inclusion criteria:

1. Informed Consent Form consistent guidelines and local legislation prior
2. Male or female patients aged at least 18 to 75 years.
3. Diagnosis of asthma according to the 2009 Global Initiative for Asthma (GINA) Guidelines.
4. Maintenance treatment with a low or medium dose of inhaled corticosteroids (ICS) with or without Long-acting beta-adrenergic (LABA), stable dose of inhaled corticosteroids (alone or in a fixed combination with a LABA) for at least for 6 weeks prior to screening.
5. Asthma control questionaire (ACQ)-6 mean score of < 1.5.
6. a. Pre-bronchodilator clinic measured FEV1 =50% and =90% of predicted normal b. FEV1 reversibility: Improvement in FEV1 =12% above baseline and an absolute change of at least 200 ml within 15-30 minutes after administration of 400 µg salbutamol.
7. Never-smokers or ex-smokers with a smoking history of less than 10 pack-years and smoking cessation at least one year prior to screening.
8. Be able to use the inhalers correctly in the opinion of the investigator.
9. Be able to perform all trial related procedures.

Exclusion criteria:

1. Significant disease other than asthma.
2. Recent history (i.e. six months or less) of myocardial infarction.
3. Hospitalisation for cardiac failure during the past year.
4. Unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
5. Lung diseases other than asthma (e.g. Chronic obstructive pulmonary disease).
6. Active tuberculosis.
7. Malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
8. Thoracotomy with pulmonary resection.
9. Alcohol or drug abuse within the past two years.
10. Pulmonary rehabilitation program
11. Hypersensitivity to LABA drugs, ciclesonide, salmeterol or any other components of the study medication delivery systems.
12. Pregnant or nursing woman.
13. Women of childbearing potential not using a highly effective method of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10

PRIMARY OUTCOMES:
FEV1 (AUC0-12h) FEV1 = Forced expiratory volume in one second, AUC = area under the curve | 12 hours

SECONDARY OUTCOMES:
FEV1 (AUC0-24h) | 24 hours
FEV1 (AUC12-24h) | 12 hours
Peak FEV1 | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1249.7.33003 Boehringer Ingelheim Investigational Site, Gières, France